CLINICAL TRIAL: NCT06637436
Title: Optimizing HIV Prevention for Highly Vulnerable Methamphetamine-using Sexual Minority Men
Brief Title: PrEP Readiness Interventions for Sustained Motivation (PRISM)
Acronym: PRISM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Adam Carrico, PhD, Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UH3AI169652 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HIV; Methamphetamine Disorders
Keywords: HIV prevention; Methamphetamine; Motivational Interviewing; Contingency Management
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (Experimental): Provides incentives for initiating PrEP care ($50) and filling a PrEP prescription ($50) in the three months following randomization.
  Interventions: Behavioral: Contingency Management (CM)
- MI+CM (Experimental): Both the CM and MI interventions described above.
  Interventions: Behavioral: Motivational Interviewing (MI); Behavioral: Contingency Management (CM)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — This telehealth MI intervention seeks to increase intrinsic motivation and self-efficacy for starting or restarting pre-exposure prophylaxis (PrEP) in session one. Session two focuses on concomitant risk behaviors such as substance use and CAS.
  Arms: MI+CM
Behavioral: Contingency Management (CM) — Provides incentives for initiating PrEP care ($50) and filling a PrEP prescription ($50) in the three months following randomization.

SUMMARY:
This is a hybrid type I, factorial randomized controlled trial to test the comparative and combined effectiveness of contingency management (CM) alone or CM with motivational interviewing (MI) for optimizing entry or re-entry into the PrEP care continuum. A total of 400 participants will be randomized to CM (n = 200) or MI+CM (n = 200), all delivered via Telehealth. Monthly follow-up assessments will be completed over 12 months to examine differential effectiveness for the primary outcome - filling a PrEP prescription (verified using a digital photo or detectable tenofovir diphosphate). Secondary outcomes will include: self-reported PrEP clinical evaluation by a PrEP provider; self-reported meth and other substance use severity (ASSIST), and self-reported receptive and insertive condomless anal sex (CAS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Assigned male a birth
* Self-reported methamphetamine use in the past 3 months
* Has not filled a PrEP prescription in the past 6 months

Exclusion Criteria:

* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Verified PrEP Use | 12 Months
  The proportion of participants providing evidence of PrEP use (i.e., a digital photo a PrEP medication bottle bearing their name, evidence of receipt of injectable PrEP from a medical record, or a dried blood spot with detectable tenofvir diphosphate for those taking daily oral PrEP)

SECONDARY OUTCOMES:
Median Time to Verified PrEP Use | 12 Months
  The number of days after randomization until evidence of PrEP use (i.e., a digital photo a PrEP medication bottle bearing their name, evidence of receipt of injectable PrEP from a medical record, or a dried blood spot with detectable tenofvir diphosphate for those taking daily oral PrEP).
Clinical Cut Points for Self-Reported Methamphetamine Use Severity | 12 Months
  Participants will complete the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), which provides validated composite scores for the severity of amphetamine and other substance use (Mild = 0-3; Moderate = 4-26; Severe = 27+).
Proportion of Participants Reporting Insertive Condomless Anal Sex (CAS) | 12 Months
  Participants will complete a detailed behavioral assessment to report the number of men with whom they have had insertive CAS in the past 3 months. Changes in the mean number of insertive CAS partners will be examined.
Proportion of Participants Reporting Receptive Condomless Anal Sex (CAS) | 12 Months
  Participants will complete a detailed behavioral assessment to report the number of men with whom they have had receptive CAS in the past 3 months. Changes in the mean number of receptive CAS partners will be examined.
Proportion of Participants with Prevention Effective PrEP Use | 12 Months
  Proportion of participants taking daily oral PrEP with tenofovir-diphosphate levels of 700 mol/punch or greater

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida International University Stempel College of Public Health and Social Work, Miami, Florida
  - Florida International University, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be uploaded to a secure database after the team completes intent-to-treat analyses of the primary and secondary outcomes.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: August 2027 (estimated start date) without an end date
Access Criteria: These data will be publicly accessible.
URL: https://www.prism-study.com